CLINICAL TRIAL: NCT06122753
Title: Transjugular Intrahepatic Portosystemic Shunt (TIPS) for Variceal Bleeding in Cirrhotic Patients With Occlusive Portal Vein Thrombosis (PVT): A Multicenter Randomized Trial
Brief Title: Preemptive TIPS for Variceal Bleeding in Cirrhotic Patients With Occlusive Portal Vein Thrombosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Beijing YouAn Hospital (Other); Beijing Friendship Hospital (Other); Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, luo xuefeng, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pTIPS-PVT
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Portal Hypertension; Portal Vein Thrombosis; Esophageal Varix Bleeding; Portosystemic Shunt
MeSH Terms: conditions — Hypertension, Portal | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Therapy (Active Comparator): Standard treatment to achieve initial hemostasis: vasoactive drugs (somatostatin or terlipressin) + endoscopic hemostasis according to the center protocol.
  Standard combined endoscopic and pharmacological therapy as secondary prophylaxis (carvedilol + repeated endoscopic variceal ligation until the eradication of the esophageal varices).
  Interventions: Procedure: standard second prophylaxis
- Preemptive TIPS (Experimental): Standard treatment to achieve initial hemostasis: vasoactive drugs (somatostatin or terlipressin) + endoscopic hemostasis according to the center protocol.
  Performance of TIPS in the first 72 hours following initial endoscopic hemostasis.
  Interventions: Procedure: preemptive TIPS

INTERVENTIONS:
Procedure: preemptive TIPS — The TIPS procedure should be performed within 72 hours after the initial endoscopic examination or treatment. An 8 mm Viatorr stent will be used for TIPS establishment. The aim will be to reduce the portal pressure gradient below 12 mm Hg. Embolization, either with coils or glue, can be performed, if it is felt necessary, especially in patients where portography shows the filling of large portosystemic collaterals feeding the varices. After TIPS, anticoagulation will not be used as a rule but is allowed if the attending physician thinks that it is warranted.
  Other Names: early TIPS
  Arms: Preemptive TIPS
Procedure: standard second prophylaxis — Patients will receive vasoactive drugs up to 5 days; then a non-selective beta-blocker (carvedilol) will be started with an initial dose of 6.25 mg, the dose of propranolol will be increased to 12.5 mg.
  The second elective session of endoscopic band ligation will be performed within the first 28 days after the initial endoscopic treatment. The following sessions will be performed at 28 +/- 3 days intervals until variceal eradication. Once eradication is achieved, endoscopic monitoring will be performed every 6 months. If varices reappear, new band ligation will be performed.
  Other Names: endoscopy plus drug treatment
  Arms: Standard Therapy

SUMMARY:
Portal vein thrombosis (PVT) can lead to a further increase in portal venous pressure and increase the risk of rebleeding. Whether patients with acute esophagogastric variceal bleeding with occlusive PVT benefit from preemptive TIPS is still controversial. The present study is directed at comparing the outcome of patients with acute variceal bleeding with occlusive PVT treated by standard therapy (vasoactive drugs + endoscopic variceal ligation) with or without preemptive TIPS (performed during the first 1-3 days after endoscopic procedure). The primary outcome is survival free of variceal rebleeding at 6 weeks from inclusion.

DETAILED DESCRIPTION:
Portal vein thrombosis (PVT) is a common complication in patients with cirrhosis, and the cumulative incidence of PVT is 4.6%, 8.2%, and 10.7% at 1 year, 3 years, and 5 years, respectively. PVT can lead to a further increase in portal venous pressure and increase the risk of rebleeding. According to Baveno VII, PVT can be classified according to the degree of occlusion of the portal trunk as complete occlusion (no continuous luminal structure), partial occlusion (≥50% thrombus obstruction of the lumen), mild occlusion (<50% thrombus obstruction of the lumen), or spongiotic degeneration (a large number of collateral vessels of the portal vein, with no visualization of the main portal vein). The results of a recent observational study suggested that patients with severe PVT with ≥50% thrombotic luminal obstruction had higher 6-week rebleeding rates (8.8% vs. 3.8%) and 1-year rebleeding rates (29.4% vs. 21.4%) after acute variceal bleeding. Our previous clinical study showed that patients with cirrhotic PVT treated with TIPS had lower rebleeding rates and significantly higher rates of portal vein recanalization, and it was inferred that patients with acute esophagogastric variceal bleeding with severe PVT might benefit from preemptive TIPS. Therefore, we propose to conduct a multicentre randomized controlled trial to enroll patients with acute esophagogastric variceal bleeding with occlusive PVT to compare the preemptive TIPS with the standardized therapy. The outcomes are rates of mortality, rebleeding, and complications.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis (diagnosed by imaging, laboratory tests, clinical symptoms, or liver biopsy);
* Admission due to acute bleeding from esophagogastric varices;
* Thrombus in the main trunk of the portal vein occupying ≥50% of the lumen.

Exclusion Criteria:

* Prior treatment with TIPS or surgical shunt;
* Presence of contraindications to endoscopic treatment, carvedilol, or TIPS;
* Presence of hepatocellular carcinoma exceeding Milan criteria;
* Presence of other systemic malignant tumors with expected survival time not exceeding 6 months;
* Presence of uncontrollable infection or sepsis;
* Presence of cardiac, pulmonary, or renal failure;
* Pregnant or lactating women;
* Refusal to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
6-week mortality | 6 weeks
  The rate of mortality during the first 6 weeks after inclusion in the study.

SECONDARY OUTCOMES:
5-day treatment failure | 5 days
  Incidence of cases requiring adjustment of treatment strategy within 5 days of initial standardised treatment: vomiting of blood or drainage of ≥100 ml of fresh blood from a gastric tube after 2 hours of treatment, hypovolemic shock, drop in haemoglobin of 30 g/L or more within 24 hours without transfusion.
1-year mortality | 1 year
  The rate of mortality during the first 1 year after inclusion in the study.
decompensation events | 1 year
  Rates with rebleeding, new overt ascites (moderate-heavy) or increased degree of ascites, overt hepatic encephalopathy (West-Heaven grades 2-4), or jaundice (total bilirubin >51 mmol/L) from 5 days after initial standardised treatment up to 1 year.
adverse events | 1 year
  Events of various complications such as infections, new tumours, organ failure, peptic ulcers, etc., occurring after randomisation up to the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Xuefeng Luo, Ph.D., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang X, Liu G, Wu J, Xiao X, Yan Y, Guo Y, Yang J, Li X, He Y, Yang L, Luo X. Small-Diameter Transjugular Intrahepatic Portosystemic Shunt versus Endoscopic Variceal Ligation Plus Propranolol for Variceal Rebleeding in Advanced Cirrhosis. Radiology. 2023 Aug;308(2):e223201. doi: 10.1148/radiol.223201. PMID 37606572
- [Result] Luo X, Wang Z, Tsauo J, Zhou B, Zhang H, Li X. Advanced Cirrhosis Combined with Portal Vein Thrombosis: A Randomized Trial of TIPS versus Endoscopic Band Ligation Plus Propranolol for the Prevention of Recurrent Esophageal Variceal Bleeding. Radiology. 2015 Jul;276(1):286-93. doi: 10.1148/radiol.15141252. Epub 2015 Mar 10. PMID 25759969